CLINICAL TRIAL: NCT01559805
Title: Efficacy Trial of a Brief Health Enhancement Intervention for Newly Diagnosed Men
Brief Title: Intervention to Improve Engagement in Care Among Newly Diagnosed HIV-positive Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAJ3106; R01MH097651 (NIH)
Record Dates: First submitted 2012-03-16; First posted 2012-03-21 (Estimated); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: HIV; Patient Compliance
Keywords: HIV; Viral Load; Risk; Patient Compliance; Homosexuality, Male; Anti-Retroviral Agents
MeSH Terms: conditions — Patient Compliance; Homosexuality, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Positive Choices (Experimental): A two-session, individually-focused intervention focusing on engagement in care, disclosure decision-making, and sexual risk reduction, with booster sessions after 1, 3 and 6 months.
  Interventions: Behavioral: Positive Choices
- Personalized Cognitive Counseling (Active Comparator): A one-session, individually-focused risk reduction intervention for MSM that has been selected by the CDC as a DEBI.
  Interventions: Behavioral: Personalized Cognitive Counseling

INTERVENTIONS:
Behavioral: Positive Choices — A two-session, individually-focused intervention focusing on engagement in care, disclosure decision-making, and sexual risk reduction, with booster sessions after 1, 3 and 6 months.
  Arms: Positive Choices
Behavioral: Personalized Cognitive Counseling — A one-session, individually-focused risk reduction intervention for MSM that has been selected by the CDC as a DEBI.
  Arms: Personalized Cognitive Counseling

SUMMARY:
The study involves delivering one of two interventions - either Promoting Action Towards Health (PATH) or Personalized Cognitive Counseling (PCC) - to 440 men who have sex with men (MSM) who have recently been diagnosed with HIV and assessing whether participants who received PATH achieve greater suppression of HIV viral load, demonstrate greater uptake of care and adherence to treatment, and engage in less sexual HIV transmission risk behavior than participants who received PCC.

* PATH consists of two preliminary sessions plus "booster" sessions after 1, 3, and 6 months.
* Personalized Cognitive Counseling consists of one session.

Participants will complete assessments before participating in their intervention (i.e., at "baseline") and at 3, 6, 9, and 12 month follow-up points. Participants' viral loads will be measured at approximately 6 and 12 months following baseline.

DETAILED DESCRIPTION:
Objectives:

The investigators will conduct a randomized controlled trial to test the efficacy of Promoting Action Towards Health (PATH), a brief health-enhancement and risk reduction intervention targeting newly HIV diagnosed men who have sex with men (MSM).

Specific Aims:

The investigators will establish the efficacy of PATH. The following hypotheses will be tested: Participants in the experimental condition will (1) achieve significantly greater suppression of HIV viral load; (2) demonstrate greater uptake of care and adherence to treatment; and (3) engage in less sexual HIV transmission risk behavior across the study duration than participants in the comparison condition.

Procedures:

440 newly HIV diagnosed (within 12 months) men will be randomly assigned to either: (1) the PATH experimental condition, or (2) the PCC comparison condition and followed for one year. HIV counselors will be trained to deliver the interventions within each condition. Assessments will be conducted at baseline, 3, 6, 9 and 12 months.

Significance:

Given increases in HIV incidence among MSM, advances in HIV treatment, and the demonstrated efficacy of early treatment in preventing HIV transmission, there is a critical need for effective interventions that can increase engagement and retention of MSM in care and reduce sexual HIV transmission risk behavior. PATH can be seamlessly integrated into medical care and translated into a sustainable model of care for newly diagnosed MSM to meet the urgent need for care programs that identify, treat, and prevent HIV infections.

ELIGIBILITY:
Inclusion Criteria:

* receiving an HIV diagnosis within the previous 12 months
* entry into HIV primary care
* residence in the greater New York metropolitan area
* aged 18 or older
* provision of written informed consent

Exclusion Criteria:

-demonstrating cognitive impairment, acute psychosis, or suicidal intent or plans

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2012-11; Primary Completion 2017-11-06 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Viral load | 12 months

SECONDARY OUTCOMES:
Sexual HIV transmission risk behavior | Baseline, post (3 months), 6, 9, and 12 months
  Timeline Followback Method (Sobell et al., 1996) for Transmission Risk Behavior, Risk Reduction Behavioral Intentions (Fisher, 1992), HIV Serostatus Disclosure (Kalichman, 2001) & HIV Disclosure or Nondisclosure (Serovich & Mosack, 2003), Risk Reduction Self-Efficacy (Kalichman, 2001), Risk Reduction Skill Enactment (Kalichman, 2001), Compulsive Sexual Behavior Inventory (Minor et al., 2007), Sexual Sensation Seeking (Kalichman & Rompa, 1995)
Care and treatment uptake/adherence | Baseline, post (3 months), 6, 9, and 12 months
  * Medical Chart/Self-report to assess Treatment Utilization
  * HIV Treatment and Risk-Related Knowledge (Kalichman, 2000)
Viral load | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick A Wilson, PhD, Principal Investigator — Columbia University; Nathan B Hansen, PhD, Principal Investigator — Yale University
Locations (4):
- United States (4):
  - Yale University, New Haven, Connecticut
  - Callen-Lorde Community Health Center, New York, New York
  - Harlem United Community AIDS Center, Inc., New York, New York
  - Mailman School of Public Health, Columbia University, New York, New York

REFERENCES:
- [Background] Sikkema KJ, Hansen NB, Kochman A, Santos J, Watt MH, Wilson PA, Delorenzo A, Laudato J, Mayer G. THE DEVELOPMENT AND FEASIBILITY OF A BRIEF RISK REDUCTION INTERVENTION FOR NEWLY HIV-DIAGNOSED MEN WHO HAVE SEX WITH MEN. J Community Psychol. 2011 Aug 1;39(6):717-732. doi: 10.1002/jcop.20463. PMID 22228917